CLINICAL TRIAL: NCT07284238
Title: Process of Configuring the Suicidal Ideation Framework: A Grounded Theory Study in Catalonia, Spain
Brief Title: Suicidal Ideation Framework: Grounded Theory Study, Catalonia
Acronym: SUIF-GT-CAT
Status: Not yet recruiting | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Sergio de la Hera Herrero, Mental Health Nurse Specialist and PhD Candidate at the Autonomous University of Barcelona (UAB), Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Other Study IDs: IIBSP-PCS-2025-176
Record Dates: First submitted 2025-11-18; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Suicide; Suicide Attempt; Suicide Ideation; Suicide Risk; Suicide Prevention
Keywords: Suicidal Ideation; Suicide; Meta-synthesis; Grounded Theory; Mental Health Nursing; High-Income Countries
MeSH Terms: conditions — Suicide; Suicide, Attempted; Suicide Prevention; Suicidal Ideation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Individuals with a history of suicide attempt: Participants aged ≥18 years residing in Catalonia who have made one or more suicide attempts within the past 6 to 36 months. They will take part in in-depth interviews or discussion groups to explore their attributed experiences related to the configuration of suicidal ideation. No clinical intervention will be delivered as part of the study. Data collection will focus on participants' narratives, contextual factors, and meaning-making processes connected to the suicide attempt and subsequent care and recovery pathways.
  Interventions: Procedure: In-Depth Qualitative Interview; Procedure: Discussion Group
- Members of their support networks: Individuals who are family members, friends, or significant others providing support to a person who has attempted suicide within the past three years. They will participate in interviews or discussion groups to describe their experiences, perceptions, and relational roles in the care, crisis management, and meaning-making processes surrounding the suicide attempt. No interventions will be administered. Data collection will focus on relational dynamics, contextual influences, and perceived barriers and facilitators in support and healthcare interactions.
  Interventions: Procedure: In-Depth Qualitative Interview; Procedure: Discussion Group
- Healthcare professionals involved in their care: Licensed healthcare professionals (e.g., mental health nurses, psychiatrists, psychologists, emergency clinicians) directly involved in the care of individuals who have attempted suicide. Participants will contribute through interviews or discussion groups exploring their clinical experiences, interpretive frameworks, and perceptions of care processes. No intervention is provided. Data collection will examine professional roles, institutional contexts, and factors shaping the configuration of suicidal ideation during assessment, treatment, and recovery trajectories.
  Interventions: Procedure: In-Depth Qualitative Interview; Procedure: Discussion Group

INTERVENTIONS:
Procedure: In-Depth Qualitative Interview — In-depth interviews aimed at exploring participants' lived experiences, meaning-making processes, and contextual factors related to the configuration of the suicidal ideation framework. Interviews will last approximately 30-45 minutes and will be conducted by the Principal Investigator in a confidential, safe, and clinically monitored setting. No clinical treatment or diagnostic procedure is administered.
Procedure: Discussion Group — Non-directive discussion groups composed of 4-6 participants from the same analytic category (suicide attempt survivors, support network members, or healthcare professionals). Sessions will last 60-90 minutes and will facilitate the collective exploration of relational, contextual, and sociocultural dynamics associated with the suicidal ideation framework. The procedure is solely qualitative and involves no therapeutic intervention or clinical manipulation.

SUMMARY:
This doctoral project aims to develop a comprehensive theoretical model of the process through which the suicidal ideation framework is configured as a symbolic, narrative, and relational expression, adopting a multiperspective approach that spans the suicide attempt and the stages of care and recovery. Moving away from biomedical reductionisms, this investigation seeks to identify shared meaning-making nuclei and discursive fractures that reflect the inherent conflictuality of the suicidal act.

Grounded in the integration of the theoretical frameworks previously outlined, this study adopts an interpretive-constructivist approach. Phase 1 will include studies conducted in OECD countries, providing a broad and conceptually diverse interpretive foundation. Phase 2, conducted in Catalonia, will deepen situated configurations, assuming that local sociocultural frameworks act as interpretive prisms for globally relevant phenomena.

Overall, this theoretical-methodological architecture not only ensures conceptual robustness and coherence, but also articulates an ethical and epistemic commitment to understanding suicide through the complexity of its human textures. By centering suffering, listening to historically silenced voices, honoring the singularity of each life trajectory, and grounding the inquiry in an ethics of care, this study aims to transcend a merely technical-instrumental logic of knowledge.

DETAILED DESCRIPTION:
Initial Analytical Premises:

It is posited that the suicidal ideation framework constitutes a symbolic, relational, dynamic, and multiperspective configuration whose emergence cannot be understood apart from the narrative, contextual, and structural arrangements mediating experiences of exclusion, hopelessness, affective disconnection, loss of vital meaning, and extreme suffering.

From this standpoint, a foundational premise is established: the suicidal ideation framework cannot be conceived as a static, universal, or univocal category. Rather, it is shaped as a constellation of meanings and signifiers in tension, woven through the interaction of ambivalences, silences, contradictions, and narrative ruptures. Such configuration emerges from complex subjective processes marked by structural inequalities, social stigma, institutional vulnerability, or care models that often render distress invisible or reduce it to pathologizing categories.

It is therefore assumed that an in-depth understanding of lived experiences attributed to the configuration process of the suicidal ideation framework-through the semiotic complexity of each perspective involved-will not only allow the identification of narrative structures and shared meaning nodes, but also help unravel discursive fractures that reflect the inherent conflictuality of the voluntary death process as a response to suffering experienced as intolerable.

Research Question:

From the perspective of individuals who have attempted suicide, members of their support networks, and healthcare professionals involved in their care-within the mental health services of the autonomous community of Catalonia, and informed by qualitative evidence from OECD countries-how is the suicidal ideation framework configured as a symbolic, narrative, and relational expression, based on the lived experiences attributed by these actors in the sociocultural and healthcare settings where they interact throughout the period encompassing the suicide attempt and the subsequent stages of care and recovery?

General Study Design:

The methodological design unfolds across two sequential and complementary phases:

* Phase 1 will adopt a qualitative systematic review methodology, using an interpretive qualitative metasynthesis design (Sandelowski & Barroso). It will integrate findings from previous qualitative and mixed-methods studies through reflexive thematic analysis (Braun & Clarke), supported by ATLAS.ti CAQDAS software. The process will follow PRISMA 2020, ENTREQ, and COREQ guidelines, selecting literature with high methodological quality (≥9/10 criteria of the JBI tool). The bibliographic search will be conducted across five international databases (PubMed, CINAHL, PsycINFO, Scopus, WoS), and screening will be performed by pairs of reviewers seeking ≥95% agreement and a Cohen's Kappa ≥0.80 to ensure inter-rater reliability.
* Phase 2 will follow an inductive qualitative methodology using a constructivist grounded theory design (Charmaz), framed within the interpretive paradigm under a relativist ontology and a subjectivist epistemology. The study population will be structured into three complementary analytical groups: (a) Individuals who have made one or more suicide attempts in the 6 months-3 years prior to the interview; (b) Members of support networks (family, friends, community); and (c) Healthcare professionals directly involved in the care of individuals who have attempted suicide. Participant recruitment will be coordinated with mental-health professionals following principles of autonomy, non-maleficence, and dignity protection. Institutional agreements will support safe referrals. Sample size will be determined by theoretical saturation. Theoretical-evolutionary sampling will be employed, and data generation techniques will include in-depth individual interviews (30-45 min) and discussion groups (4-6 participants, 60-90 min). Sessions will be conducted in authorised hospital or community settings, with an observer noting field data. Qualitative material, collected through audio recording, will undergo inductive-interpretive qualitative content analysis informed by constructivist grounded theory: initial coding, focused coding, and theoretical integration. An abductive logic will guide movement between data and conceptualisation. Constant comparison, analytic memos, conceptual diagrams, and conditional matrices will ensure rigour. Triangulation, participant-involvement workshops, and external audit will strengthen quality. ATLAS.ti will support systematic data management. Data handling will follow the Declaration of Helsinki and GDPR. The PI is responsible for database creation and integrity.

Phase 1 Biases and Limitations:

Publication bias: mitigated through inclusion of qualitative systematic reviews and critical heterogeneity analysis.

Language limitation: mitigated through inclusion of multicentric studies and triangulation with technical/institutional reports.

Phase 2 Biases and Limitations:

Researcher bias: mitigated through reflexivity, peer review, constant comparison, and participant validation.

Selection bias: mitigated through diverse theoretical sampling and safe inclusion of vulnerable profiles.

Participant response bias: mitigated through emotionally safe environments, rapport, neutral questioning, and professional accompaniment when needed.

Quality Control:

The PI will ensure accuracy and consistency in the Case Report Forms, maintain documentation for ≥10 years, and provide access to monitors, auditors, ethics committees, and regulatory authorities upon request.

Conclusion:

This innovative interpretive contribution represents an ethical commitment to restoring the agency of the actors involved. Ultimately, this research proposal acknowledges the role of the nursing profession as an operative agent of change and as a privileged epistemic subject in confronting one of the most complex and silenced phenomena of contemporary human experience.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age.
* Usual residence in Catalonia (Spain).
* Ability to understand, speak, read, and write in Catalan or Spanish.
* Belonging to one of the three defined analytical groups:

(A) Individuals who have attempted suicide within the past 6 months to 3 years. (B) Members of their family, social, or community support networks. (C) Healthcare professionals directly involved in the care of individuals who have attempted suicide.

* Demonstrated clinical/emotional stability ensuring safe participation, as confirmed by the referring clinician.
* For individuals with lived experience (Group A): at least 6 months since the last suicide attempt or acute clinical crisis.
* For support networks (Group B): having maintained meaningful proximity or involvement during or after the suicide attempt.
* For healthcare professionals (Group C): minimum of 1 year of professional experience in mental health care.

Exclusion Criteria:

* Presence of acute clinical decompensation preventing safe participation.
* Active suicidal risk or acute crisis at the time of recruitment.
* Acute vulnerability identified during screening.
* Inability to provide informed consent.
* Direct hierarchical dependence or conflict of interest with the research team (for Group C).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises three analytically complementary groups within the mental health system of Catalonia: (1) adults with a history of one or more suicide attempts within the past 6 months to 3 years; (2) members of their family, social, or community support networks who have provided meaningful accompaniment during or after the attempt; and (3) healthcare professionals directly involved in the care of individuals who have attempted suicide and with at least one year of experience in mental health services.
  These groups are independent from each other, ensuring contextual diversity, confidentiality and robust interpretive depth.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Conceptual Synthesis of Qualitative Findings. | Through Phase 1 completion, an average of 12-18 months.
  Generation of a third-order conceptual synthesis integrating first- and second-order findings from qualitative and mixed-methods studies conducted in OECD countries. This synthesis will be developed through reflexive thematic analysis and will provide a high-order interpretative framework that will:
  1. consolidate cross-contextual patterns and divergences in experiences attributed to suicide.
  2. inform the initial theoretical orientation of Phase 2.
  3. guide purposive and theoretical sampling.
  4. support the development of initial coding strategies in the constructivist grounded theory phase.
  Measure Type: Qualitative interpretative meta-synthesis conceptual output.
Emergent Theoretical Model. | Through study completion, an average of 24-30 months.
  Qualitative identification, comparative analysis and inductive-interpretive integration of the main categories, subcategories and theoretical relationships that explain how the suicidal ideation framework is configured as a symbolic, narrative and relational phenomenon. This outcome captures the core theoretical structure produced through initial coding, focused coding and theoretical integration, derived from the constructivist grounded theory analysis of interviews and discussion groups.
  Measure Type: Qualitative conceptual model (Grounded Theory).

SECONDARY OUTCOMES:
Identified Narrative Structures and Meaning-Making Patterns. | Through study completion, an average of 24-30 months.
  Qualitative identification of narrative structures, ambivalences, silences, contradictions and discursive ruptures attributed by participants to the process of configuring the suicidal ideation framework, across the three analytic groups (individuals with suicide attempt history, members of support networks, healthcare professionals).
  Measure Type: Qualitative thematic patterns (Reflexive Thematic Analysis).
Influence of Socio-cultural and Biographical Factors. | Through study completion, an average of 24-30 months.
  Inductive analysis of how socioaffective bonds, sociocultural frames, structural inequalities and biographical trajectories shape and modulate the subjective and relational processes involved in the configuration of the suicidal ideation framework.
  Measure Type: Qualitative thematic and relational patterns.
Relational and Contextual Mechanisms. | Through study completion, an average of 24-30 months.
  Examination of how relational dynamics, contextual interactions and social environments contribute to modelling the configuration of the suicidal ideation framework across different participant groups.
  Measure Type: Qualitative category development.
Perceived Barriers and Facilitators in Healthcare. | Through study completion, an average of 24-30 months.
  Identification of perceived barriers, facilitators, protective factors and contextual conditions present in mental health and emergency care settings, as described by individuals with suicide attempt history, their support networks and healthcare professionals.
  Measure Type: Qualitative thematic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Sergio de la Hera Herrero, Bachelor of Science in Nursing, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared. This is a qualitative study involving highly sensitive narratives related to suicide attempts, emotional distress, and personal life histories. In accordance with ethical requirements of the Comitè d'Ètica d'Investigació amb Medicaments de l'Hospital de la Santa Creu i Sant Pau (CEIm-Sant Pau), the informed consent agreement, and the EU General Data Protection Regulation (GDPR), the IPD cannot be made available to external researchers because re-identification cannot be fully prevented even after de-identification or pseudonymization.
  However, the study will make available:
  * Aggregated thematic findings
  * Category structures
  * Coding frameworks
  * The final substantive grounded theory model
  * The third-order interpretative synthesis (Phase 1)
  These outputs may be shared upon reasonable request in compliance with all regulatory and ethical safeguards.

REFERENCES:
- [Background] Union Européenne. Regulation (EU) 2016/679 of the European Parliament and of the Council of 27 April 2016 (General Data Protection Regulation). Off J Eur Union. 2016;L119:1-88.
- [Background] McHugh ML. Interrater reliability: the kappa statistic. Biochem Med (Zagreb). 2012;22(3):276-82. PMID 23092060
- [Background] Aromataris E, Munn Z, editors. JBI Manual for Evidence Synthesis. Adelaide: Joanna Briggs Institute; 2020.
- [Background] Tong A, Sainsbury P, Craig J. Consolidated criteria for reporting qualitative research (COREQ): a 32-item checklist for interviews and focus groups. Int J Qual Health Care. 2007 Dec;19(6):349-57. doi: 10.1093/intqhc/mzm042. Epub 2007 Sep 14. PMID 17872937
- [Background] Tong A, Flemming K, McInnes E, Oliver S, Craig J. Enhancing transparency in reporting the synthesis of qualitative research: ENTREQ. BMC Med Res Methodol. 2012 Nov 27;12:181. doi: 10.1186/1471-2288-12-181. PMID 23185978
- [Background] Page MJ, McKenzie JE, Bossuyt PM, Boutron I, Hoffmann TC, Mulrow CD, Shamseer L, Tetzlaff JM, Akl EA, Brennan SE, Chou R, Glanville J, Grimshaw JM, Hrobjartsson A, Lalu MM, Li T, Loder EW, Mayo-Wilson E, McDonald S, McGuinness LA, Stewart LA, Thomas J, Tricco AC, Welch VA, Whiting P, Moher D. The PRISMA 2020 statement: an updated guideline for reporting systematic reviews. BMJ. 2021 Mar 29;372:n71. doi: 10.1136/bmj.n71. PMID 33782057
- [Background] Charmaz K. Constructing grounded theory. 2nd ed. Thousand Oaks: Sage; 2014.
- [Background] Strauss A, Corbin J. Basics of qualitative research: Techniques and procedures for developing grounded theory. 2nd ed. Thousand Oaks: Sage; 1998.
- [Background] Braun V, Clarke V. Using thematic analysis in psychology. Qual Res Psychol. 2006;3(2):77-101.
- [Background] Sandelowski M, Barroso J. Handbook for synthesizing qualitative research. New York: Springer; 2007.
- [Background] Ministerio de Sanidad. Estrategia de Salud Mental del Sistema Nacional de Salud 2022-2026. Madrid: Ministerio de Sanidad; 2022.Aromataris E, Munn Z, editors. JBI Manual for Evidence Synthesis. JBI; 2020.
- [Background] Talseth AG, Gilje F, Norberg A. The significance of meaningful and confirming relationships as protective factors in suicidal patients: a qualitative study. Scand J Caring Sci. 2001;15(4):257-64.
- [Background] Cutcliffe JR, Santos JC. Involving individuals who have experienced suicide: a call to action. Issues Ment Health Nurs. 2012;33(4):244-8.
- [Background] Kral MJ. Suicide and the transformation of identity: A psychosocial approach. In: White J, Marsh IB, Kral MJ, Morris J, editors. Critical Suicidology. Vancouver: UBC Press; 2016. p. 71-87.
- [Background] McAdams DP. The stories we live by: Personal myths and the making of the self. New York: The Guilford Press; 1993.
- [Background] Hjelmeland H, Knizek BL. Why we need qualitative research in suicidology. Suicide Life Threat Behav. 2010 Feb;40(1):74-80. doi: 10.1521/suli.2010.40.1.74. PMID 20170263
- [Background] Sun FK, Long A, Boore J. The attitudes of casualty nurses in Taiwan to patients who have attempted suicide. J Clin Nurs. 2007 Feb;16(2):255-63. doi: 10.1111/j.1365-2702.2005.01479.x. PMID 17239060
- [Background] Talseth AG, Gilje F, Norberg A. Being met - a passageway to hope for relatives of suicidal people: A hermeneutic perspective. Perspect Psychiatr Care. 2003;39(2):61-70.
- [Background] Cutcliffe JR. The differences and commonalities between United Kingdom and Canadian Psychiatric/Mental Health nursing: a personal reflection. J Psychiatr Ment Health Nurs. 2003 Jun;10(3):255-7. doi: 10.1046/j.1365-2850.2003.00637.x. No abstract available. PMID 12755909
- [Background] Travelbee J. Interpersonal aspects of nursing. Philadelphia: FA Davis Company; 1971.
- [Background] Shneidman ES. The psychache: A clinical approach to suicide. Northvale (NJ): Jason Aronson; 1993.
- [Background] Klonsky ED, May AM. The three-step theory (3ST): A new theory of suicide rooted in the "ideation-to-action" framework. Int J Cogn Ther. 2015;8(2):114-29.
- [Background] O'Connor RC, Kirtley OJ. The integrated motivational-volitional model of suicidal behaviour. Philos Trans R Soc Lond B Biol Sci. 2018 Sep 5;373(1754):20170268. doi: 10.1098/rstb.2017.0268. PMID 30012735
- [Background] Kleinman A. Social suffering. Berkeley: University of California Press; 1997.
- [Background] Durkheim E. Le suicide: Étude de sociologie. Paris: Félix Alcan; 1897.
- [Background] White J, Marsh IB, Kral MJ, Morris J. Critical Suicidology: Transforming Suicide Research and Prevention for the 21st Century. Vancouver: UBC Press; 2016.
- [Background] Fitzpatrick SJ. Understanding suicide as social suffering: A review of recent social work literature. Health Soc Work. 2018;43(4):219-27.
- [Background] Chandler A. Youth suicide and the politics of silence: Reflections on research practice. Crit Public Health. 2019;29(2):140-50.
- See also: Registered protocol for the qualitative meta-synthesis (Phase 1) in PROSPERO-CRD420251036324 — https://www.crd.york.ac.uk/PROSPERO/view/CRD420251036324
- See also: Full preregistered study protocol and supplementary methodological materials hosted on the Open Science Framework (OSF). — https://doi.org/10.17605/OSF.IO/AWXVP